CLINICAL TRIAL: NCT05542329
Title: Efficiency of a Telemedicine-based Follow-up on for the Medical Management of Patients Leaving the Intensive Care Unit
Acronym: TéléRéa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8940
Record Dates: First submitted 2022-09-09; First posted 2022-09-15 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Care After Going to Intensive Care
Keywords: Tele-medicine; Intensive Care Unit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of care
- Tele-Medecine (Experimental): The experimental group will be given a case of connected devices dedicated to telemedicine allowing them to closely monitor their state of health during the 3 months following discharge from hospital
  Interventions: Device: Monitoring by Tele-Medecine

INTERVENTIONS:
Device: Monitoring by Tele-Medecine — Monitoring by Tele-Medecine
  Arms: Tele-Medecine

SUMMARY:
Patients surviving to a stay in intensive care unit (ICU) are likely to require specific care and follow-up after their ICU stay, in order to manage the serious illness at the origin of the ICU stay and any sequelae, but also to adapt the treatments and prevent new complications. At present, there is no specific care chain after ICU.

In order to meet this need, we propose the implementation of a care chain integrating telemedicine at home. We compare the current system (lack of specific follow-up) to follow-up by telemedicine at home.

ELIGIBILITY:
Inclusion criteria:

* Adult patient ≥ 18 years old
* Patient admitted to ICU
* Stay in intensive care > 48h
* Patient having benefited from at least one organ support during the ICU stay: invasive or non-invasive ventilation (including nasal high-flow oxygen therapy), inotropic or vasopressor support, renal replacement therapy)
* Understanding of the French language
* Patient or entourage able to carry out the measures proposed by telemedicine
* Subject affiliated to a social health insurance scheme
* Subject having signed a consent form

Exclusion criteria:

* Subject under guardianship or curatorship
* Pregnancy / lactation
* Voluntary drug poisoning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the medico-economic of telemedicine monitoring | 12 month
  The main judgment criterion will be the incremental cost-utility ratio of the innovation represented by monitoring by a telemedicine device linked to a nurse coordination unit, compared to the usual monitoring without telemedicine.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Service de Réanimation Médicale - CH Dijon, Dijon
  - Service de Réanimation Médicale - CH Mulhouse, Mulhouse
  - Service de Réanimation Médicale - CHRU Nancy - France, Nancy
  - Service de Médecine Intensive - Réanimation / CHU Strasbourg - France, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided